CLINICAL TRIAL: NCT05082142
Title: Tranexamic Acid to Improve Same-day Discharge Rates After Holmium Laser Enucleation of the Prostate (HoLEP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Professor of Urology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00215134
Record Dates: First submitted 2021-09-24; First posted 2021-10-18 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Kidney Calculi; Urologic Diseases; Benign Prostatic Hypertrophy
MeSH Terms: conditions — Kidney Calculi; Urologic Diseases; Prostatic Hyperplasia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TXA intraoperatively (Experimental): Patients will receive intraoperative 1g TXA during the HoLEP procedure.
  Interventions: Drug: Tranexamic acid
- No TXA intraoperatively (No Intervention): Patients will not receive intraoperative TXA during the HoLEP procedure.

INTERVENTIONS:
Drug: Tranexamic acid — Patients in the intervention arm will receive 1g of intraoperative IV TXA during the HoLEP procedure.
  Arms: TXA intraoperatively

SUMMARY:
This study is designed to assess if there is a significant difference in same day discharge rates after Holmium Laser Enucleation of the Prostate (HoLEP). The investigators attempt to perform HoLEP as a same-day discharge (SDD) procedure, but at Northwestern Memorial, the SDD rate is currently approximately 60%. The limiting factor in SDD is hematuria. Tranexamic acid (TXA) is a clot promoting drug that is commonly used by orthopedic, cardiac and obstetric surgeons to prevent bleeding. The primary outcome will be to assess if there is a difference in SDD rates in those who receive TXA vs. those who do not.

Secondary outcomes will assess bleeding complications (defined as unplanned ED visit/clinic visit/procedure/admission related to bleeding, clot retention, clot evacuation, need for perioperative transfusion) between participants who receive TXA vs. those do not. The study will also assess differences in perioperative complications associated with TXA including but not limited to: deep venous thrombosis, pulmonary embolism, cerebrovascular events, between the groups. The study will also assess for the duration of postoperative hematuria between groups as well as differences in operative times between the groups.

The investigators anticipate that there may be up to a 25% increase in SDD rates in those who receive TXA vs. those who do not.

DETAILED DESCRIPTION:
On the day of the surgery, the treatment assigned to the participant will be determined by chance, like flipping a coin. One arm will undergo the HoLEP procedure while receiving 1g TXA IV intraoperatively. The second arm will undergo the HoLEP procedure without receiving TXA IV intraoperatively.

After surgery, participants will receive weekly surveys via text message or email asking them to report any instances of difficulty urinating or blood in the urine. These surveys will continue for 12 weeks.

30 days after surgery, participants will come in for a standard clinical follow up appointment where they will be asked to complete a questionnaire about bleeding complications and symptoms.

12 weeks after surgery, participants will come in for their 12-week follow up and will be assessed for benign prostate hyperplasia (BPH) symptoms and their urine flow rate will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Males 18-89 undergoing HoLEP
* Willing to sign the Informed Consent Form
* Able to read, understand, and complete patient questionnaires, pain texts, and medication diary

Exclusion Criteria:

* Allergy or hypersensitivity to TXA, history of acute venous or arterial thrombosis, intrinsic risk for thrombosis or thromboembolism, history of thromboembolic disease, hereditary thrombophilia, use of hormonal agents
* Patients having any additional simultaneous procedure other than a HoLEP (cystolitholapaxy allowed).
* Anticipated need for perineal urethrostomy at the time of HoLEP
* Patient not undergoing catheter removal and voiding trial at Northwestern Memorial Hospital

Ages: 18 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Assmus MA, Lee MS, Helon JW, Krambeck AE. Tranexamic Acid Does Not Improve Outcomes of Holmium Laser Enucleation of the Prostate: A Prospective Randomized Controlled Trial. J Endourol. 2023 Feb;37(2):171-178. doi: 10.1089/end.2022.0407. Epub 2022 Dec 27. PMID 36222618

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Median (Full Range); unit: years] | 69.1 [56 to 87.1] | 69.7 [52.1 to 87.6] | 69.4 [52.1 to 87.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 55 | 55 | 110
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55 | 55 | 110
Pre-op Prostate size, continious [Median (Full Range); unit: cc] | 114 [73 to 150] | 105.5 [76.8 to 128.3] | 109.8 [73 to 150]

OUTCOME MEASURES:

1. Primary Outcome: Same-day Discharge Rate
Description: Number of participants who are discharged on the same day and have same-day catheter removal.
Time Frame: Day 0-1
Measure: Count of Participants; unit: Participants
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
Number analyzed (Participants) | 55 | 55
Participants | 50 | 49

2. Primary Outcome: Length of Stay
Description: Post-operative to discharge home
Time Frame: Day 0-1
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
Number analyzed (Participants) | 55 | 55
minutes | 170 [127 to 243] | 187 [141 to 320]

3. Primary Outcome: Same Day Discharge
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
Number analyzed (Participants) | 55 | 55
Participants | 51 | 49

4. Secondary Outcome: Number of Participants With Bleeding Complications
Description: Participants who have bleeding complications (defined as unplanned ED visit/clinic/procedure/admission related to bleeding, clot retention, clot evacuation, need for perioperative transfusion). This will be assessed by a weekly survey distributed to participants for 12 weeks.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
Number analyzed (Participants) | 55 | 55
Participants | 4 | 6

5. Secondary Outcome: Duration of Postoperative Hematuria
Description: Days participants have postoperative hematuria. This will be assessed by a weekly survey distributed to participants for 12 weeks.
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Operative Times
Description: Operative times during HoLEP procedure.
Time Frame: Day 0
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
Number analyzed (Participants) | 55 | 55
minutes | 58 [46.5 to 75.5] | 53 [43 to 70.5]

7. Secondary Outcome: Adverse Events Related to TXA
Description: Number of participants who have adverse events related to TXA (thrombotic events (DVT, PE, stroke), seizures).
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
Number analyzed (Participants) | 55 | 55
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 90-day complications post-operatively
Description: Clavien Dindo classification was used to categorize complications
Arm/Group | TXA Intraoperatively | No TXA Intraoperatively
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 1/55 | 0/55
Other Adverse Events (participants affected / at risk) | 9/55 | 17/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXA Intraoperatively (N=55) | No TXA Intraoperatively (N=55)
CD IIIb (Renal and urinary disorders) | 1 (1) | 0 (0) — ureteroscopy for obstructing ureteral stone
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXA Intraoperatively (N=55) | No TXA Intraoperatively (N=55)
CD I (Renal and urinary disorders) | 7 (55) | 15 (55)
CD II (Renal and urinary disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05082142/Prot_002.pdf
  • Informed Consent Form (2021-10-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT05082142/ICF_001.pdf